CLINICAL TRIAL: NCT02293941
Title: A Phase 2, Randomized, Multiple-dose, Double-blind, Placebo-controlled Study of JKB-122 to Assess Liver Tests in HCV Subjects Who Have Been Nonresponsive to Prior Interferon Based Therapies Either Alone or in Combination With Ribavirin
Brief Title: Liver Test Study of Using JKB-122 in Hepatitis C Virus (HCV)-Positive Patients Nonresponsive to Prior Interferon Based Therapies
Acronym: JKB122
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Completed stage I without pursuing stage II
Sponsor: TaiwanJ Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JKB122; NCT02149368 (obsolete NCT alias)
Record Dates: First submitted 2014-11-13; First posted 2014-11-19 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Chronic Hepatitis C
Keywords: liver inflammation
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis | interventions — JKB-122

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- JKB-122 5mg (Experimental): 5mg, oral, once daily
  Interventions: Drug: JKB-122 5mg
- JKB-122 15 mg (Experimental): 15mg, oral, once daily
  Interventions: Drug: JKB-122 15mg
- JKB-122 35 mg (Experimental): 35mg, oral, once daily
  Interventions: Drug: JKB-122 35mg
- placebo (Placebo Comparator): comparable capsule, oral, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JKB-122 5mg — Participants were randomized to receive JKB-122 5mg for 12 weeks
  Arms: JKB-122 5mg
Drug: JKB-122 15mg — Participants were randomized to receive JKB-122 15mg for 12 weeks
  Arms: JKB-122 15 mg
Drug: JKB-122 35mg — Participants were randomized to receive JKB-122 35mg for 12 weeks
  Arms: JKB-122 35 mg
Drug: Placebo — Participants were randomized to receive comparable placebo for 12 weeks
  Arms: placebo

SUMMARY:
The primary objective of this study is to assess changes in alanine aminotransferase (ALT) in hepatitis C virus (HCV)-infected subjects given daily doses of JKB-122 for 3 months who have been nonresponsive to, intolerable to, or relapsed from prior interferon-based therapies (pegylated or standard) either alone or in combination with ribavirin or other anti-HCV therapies including direct-acting anti-viral agents.

ELIGIBILITY:
Inclusion Criteria:

* Is HCV positive (documented by HCV RNA testing at Screening). Chronic hepatitis C is defined as a) Positive for anti-HCV antibody, HCV RNA, or an HCV genotype at least 6 months before screening, and positive for HCV RNA and anti-HCV antibody at the time of screening; or b) Positive for anti-HCV antibody and HCV RNA at the time of screening with a liver biopsy consistent with chronic HCV infection (or a liver biopsy performed before enrollment with evidence of CHC disease, such as the presence of fibrosis), according to "Guidance for Industry. Chronic Hepatitis C Virus Infection: Developing Direct-Acting Antiviral Agents for Treatment".
* Has previous results from HCV genotype testing. If previous results are not available, such testing should be performed at Screening.
* Has had a liver biopsy or Fibroscan™ within 3 years and the severity of hepatic dysfunction is limited to the following:

  * Metavir Stage 0 to stage 3 fibrosis (according to liver biopsy) or Fibroscan™ results
  * ALT and AST values not exceeding 5 x ULN (Baseline value for each parameter will be calculated as the average of 3 values obtained 7 days apart
  * Normal total bilirubin, and prothrombin time/INR values
* Has elevated liver test results (ALT) at least 1.5 x ULN and not exceeding 5 x ULN (Baseline value for each parameter will be calculated as the average of 3 values obtained 7 days apart
* Is refractory or null responder, intolerable, relapser, or partial responder.

  * Null responder is defined as less than a 2 log10 IU/mL reduction in HCV RNA after 12 weeks of treatment with standard or Peg Interferon/ribavirin or other anti-HCV therapies;
  * Relapser is defined as HCV RNA undetectable (or negative, per site's definition) at the end stage of treatment with a standard or pegylated interferon-based regimen or other anti-HCV therapies, but HCV RNA detectable during post-treatment follow-up;
  * The intolerable is defined as HCV patients who cannot tolerate the side effects of previous interferon-based therapies or other anti-HCV therapies, or who were not suitable for interferon-based therapies or other anti-HCV therapies;
  * Partial responder is defined as achieved more than 2 log10 IU/mL reduction in HCV RNA by Week 12 (± 1 week) during a prior pegIFN/RBV treatment course or other anti-HCV therapies but failed to achieve HCV RNA undetectable at the end stage of treatment.

Exclusion Criteria:

1. Has history of allergy to JKB-122 or related compounds
2. Has human immunodeficiency virus (HIV) or is hepatitis B positive
3. Is with a current diagnosis of cirrhosis, both compensated and uncompensated Child-Pugh A, B or C
4. Has positive urine drug screen at Screening
5. Is currently consuming greater than 30 g of alcohol per day (eg, 2 highballs with 1 shot each, or 2 beers) or has consumed greater than 2 glasses of alcohol per day within 3 months prior to the first screening visit (Day -28)
6. Is being treated with any prescription narcotic drug (including transdermal delivery systems)
7. Has a known or suspected central nervous system disorder that may predispose to seizures or lower the seizure threshold
8. Has unstable and uncontrollable hypertension (>180/110 mmHg)
9. Has received other therapies for HCV infection (interferon, pegylated interferon, ribavirin, or others) in the last 4 weeks prior to the first screening visit (Day -28)
10. Requires concomitant use of or treatment with opioids or other excluded drugs such as hepatotoxic medications
11. Has received other investigational agents within 30 days prior to the first screening visit (Day -28)
12. Has a disease that would require chronic use of prescription corticosteroids
13. Has either autoimmune or genetic liver disease
14. May be chronically or latently infected with microbial agents other than HCV
15. Has impaired renal function
16. Has BMI> 30 or BMI <18
17. If female, pregnant or lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-05; Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
ALT | baseline and 12 weeks
  To assess changes in ALT in HCV-infected subjects given daily doses of JKB-122

SECONDARY OUTCOMES:
Pharmacokinetic analysis (plasma concentration of JKB-122) | Day 1, 29, 57, 78
  plasma concentration of JKB-122 will be measured for exploration of exposure/response relationships in all subjects of each dose group at Stage 1.
Clinical laboratory tests (Includes hematology, coagulation, and serum chemistry.) | Screening, Day 1, 15, 29, 57, 85 and 30 days after EOS
  Includes hematology, coagulation, and serum chemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Chu Shih, PhD, Study Director — TaiwanJ Pharmaceuticals
Locations (14):
- Taiwan (14):
  - Changhua Christian Hospital, Changhua
  - Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Chiayi City
  - Chang Gung Memorial Hospital, Chiayi, Chiayi City
  - Chia-Yi Christian Hospital, Chiayi City
  - Chang Gung Memorial Hospital, Kaohsiung, Kaohsiung City
  - Chang Gung Memorial Hospital, Keelung, Keelung
  - Chi Mei Medical Center - Liouying Branch, Tainan
  - Chi Mei Hospital, YongKang Branch, Tainan
  - Cathay General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
  - China Medical University Beigang Hospital, Yuanlin
  - National Taiwan University Hospital, Yun-Lin Branch, Yuanlin